CLINICAL TRIAL: NCT06037733
Title: Primary Tumor Radiotherapy Omitting Clinical Target Volume for Patients With Advanced Non Small Cell Lung Cancer Responded to Immunotherapy and Chemotherapy
Brief Title: Primary Tumor Radiotherapy Omitting CTV for Patients With Advanced NSCLC Responded to Immunotherapy and Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, Director of the department of Radiotherapy Oncology, Hubei Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OMCTV-HC-002
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Advanced Non-Small Cell Squamous Lung Cancer; Radiotherapy; Immunotherapy
Keywords: omitting CTV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTV-omitted (Experimental): CTV was omitted for primary tumor radiotherapy for advanced NSCLC who responded to therapy with immunotherapy and chemotherapy.
  Interventions: Radiation: CTV omitted or delineated
- CTV-delineated (Active Comparator): CTV was delineated for primary tumor radiotherapy for advanced NSCLC who responded to induction therapy with immunotherapy and chemotherapy.
  Interventions: Radiation: CTV omitted or delineated

INTERVENTIONS:
Radiation: CTV omitted or delineated — Patients who responded to the therapy (immunotherapy and chemotherapy) were randomly (1:1) assigned into CTV-omitted radiotherapy group or CTV-delineated radiotherapy group.

SUMMARY:
The aim of this randomized study is to investigate pneumonitis, local tumor control, and survival outcomes of primary tumor radiotherapy omitting CTV for patients with advanced NSCLC responded to immunotherapy and chemotherapy

DETAILED DESCRIPTION:
Studies have confirmed that systemic therapy combined with primary tumor radiotherapy can improve symptoms and prolong survival of advanced NSCLC. Our previous sturdy indicated that patients who received immunotherapy and subsequent radiotherapy suffered higher proportion of pneumonitis. Patients suffered grade 2 or more pneumonitis have worse prognosis. It is urged to optimize the radiotherapy dose and target volume for patients treated with immunotherapy and radiotherapy. According to retrospective and prospective studies, omitting primary tumor CTV radiation therapy showed no reduction in local control and survival for locally advanced NSCLC. It is postulated that omitting CTV radiation for patients responded to therapy with immunotherapy and chemotherapy will have less pneumonitis without sacrificing the local control rate. Omitting CTV may also retain better immune function which will facilitate the immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced non-small cell lung cancer (according to the 8th edition of the TNM cancer staging system of AJCC and UICC);
2. After over two cycles of chemotherapy combined with immunotherapy, the efficacy was CR, PR or SD (with a decreasing trend);
3. Age 18 to 80 years old, performance status 0-1;
4. measurable or evaluable lesions;
5. Survival expectancy is not less than 6 months;
6. adequate cardiac, pulmonary, renal, and hepatic and bone marrow function

Exclusion Criteria:

1. tumor progress after therapy with immunotherapy and chemotherapy
2. EGFR, ALK, or ROS1 mutation;
3. Previous thoracic radiotherapy;
4. grade 2 or more immune-related adverse events after induction immunotherapy
5. Previous malignancies (except stage I non-melanic skin cancer or cervical carcinoma in situ);
6. Pregnant or lactating women
7. undergoing other clinical trials;
8. Have serious comorbidities, including myocardial infarction, severe arrhythmia, severe cerebrovascular disease, ulcer disease, psychosis and uncontrollable diabetes;
9. Patients with HIV positive and undergoing antiviral therapy;
10. Active tuberculosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-03-13 (Estimated); Primary Completion 2026-03-13 (Estimated); Study Completion 2027-10-08 (Estimated)

PRIMARY OUTCOMES:
grade 2 or more pneumonitis | up to 6 months

SECONDARY OUTCOMES:
local/regional control rate | up to 12 months
Progress free survival | up to 12 months
grade 3 or more pneumonitis | up to 6 months
grade 3 or more esophagitis | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guang Han, PhD, Principal Investigator — Department of Radiation Oncology, Hubei Cancer Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China